CLINICAL TRIAL: NCT06901921
Title: Responsiveness and Minimal Clinically Important Difference (MCID) of Knee Injury and Osteoarthritis Outcome Score-12 (KOOS-12) in Patients With Knee Osteoarthritis (OA): A Prospective Cohort Study.
Brief Title: Responsiveness and Minimal Clinically Important Difference (MCID) of Knee Injury and Osteoarthritis (KOOS-12) in (OA)
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/780
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PT-intervention
  Interventions: Diagnostic Test: PT-intervention

INTERVENTIONS:
Diagnostic Test: PT-intervention — 60 participants undergoing PT-intervention for about 3 months will be taken and questionnaire (KOOS-12) will be filled by them at regular intervals of baseline, 4, 8 and 12 weeks respectively while global rating of change questionnaire will be filled by them at start and end of intervention and these values will be compared to see if patients' condition has improved or not.

SUMMARY:
Osteoarthritis (OA) is a common and disabling constant Musculoskeletal Disorder that causes significant weight on individual, Health Care Systems, and social economy. With the maturing of the populace and the commonness of undesirable way of life practices, the predominance and disease burden of OA are expanding day by day. Different non-surgical interventions have been introduced worldwide for the treatment of knee OA. The aim of this study is to determine the responsiveness and minimal clinically important difference for knee injury and osteoarthritis outcome score-12 in knee OA patients respectively.

ELIGIBILITY:
Inclusion Criteria:

* An Age group of 50-65 years will be included in study.
* both males and females will be included.
* Patients with Unilateral knee OA with K-L grade II-III involving medial side will be a part of study.
* Following ACR (American college of rheumatology) guidelines Patient with knee pain must have 3 or more than 3 of the following symptoms i.e. age >50 years, morning stiffness <30 minutes, crepitus on movement, tenderness, bony enlargements, no palpable warmth will also be a part of study.
* patient having pain ranging from 5-8 on Numeral Pain Rating Scale (NPRS) will be included

Exclusion Criteria:

* participants with Traumatic knee injuries (cruciate injuries, meniscal injuries etc.) will be excluded.
* Osteonecrosis patients will be excluded.
* Patient with Neurological problems won't be a part of this study.
* People having Metastasis or neoplasm will be omitted.
* Knee or hip fractures
* Rheumatoid arthritis, Systemic lupus erythematosus (SLE) or other autoimmune disease people will be listed out.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoarthritis (OA) is a common and disabling constant Musculoskeletal Disorder that causes significant weight on individual, Health Care Systems, and social economy. With the maturing of the populace and the commonness of undesirable way of life practices, the predominance and disease burden of OA are expanding day by day. Different non-surgical interventions have been introduced worldwide for the treatment of knee OA. The aim of this study is to determine the responsiveness and minimal clinically important difference for knee injury and osteoarthritis outcome score-12 in knee OA patients respectively.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Knee injury and osteoarthritis outcome score-12 (KOOS-12) | 12 Months
  It mainly consisted of 3 sub-parts having 12 questions that include Pain, Function, and QOL. No. of score for each item is from 0-4 and the mean score is 100 where 0 indicates dangerous practical difficulties and 100 indicates normality.
  Scale Name:2.2.
GLOBAL RATING OF CHANGE (GRC) USING ANCHOR-BASED METHOD | 12 months
  This questionnaire will ask the participators to evaluate their present condition with their baseline condition. The scale consists of 15 points on it from -7 to 7, whereby -7 displays a very great deal worse, 0 symbols as remain same, and 7 reflects as a very great deal better. This is used to classify the members into the "change" group including points ±6-±7 points and "no change" group including 0-±5 points for evaluating MCID.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No